CLINICAL TRIAL: NCT03407937
Title: The Role of the Endocannabinoids During the Analgesia Caused by Hypnosis and Meditation
Brief Title: The Effect of Hypnosis on Blood Concentrations of Endocannabinoids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-1477
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2017-10

CONDITIONS: Hypnosis; Endocannabinoids; Analgesia
Keywords: Hypnosis; Meditation; Conditioned pain modulation; Placebo; Endocannabinoids; Opioid peptides; Norepinephrine; Pain; Analgesia; Genes; Heart rate variability
MeSH Terms: conditions — Agnosia; Pain | interventions — Hypnosis; Meditation; Mindfulness; Diffuse Noxious Inhibitory Control; Placebo Effect

STUDY DESIGN:
Intervention Model Description: Repeated measures on a single group of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Receiving the conditioned pain modulation intervention during the first session and receiving the placebo and the hypnosis or meditation interventions during the second session.
  Interventions: Behavioral: Hypnosis; Behavioral: Meditation; Other: Conditioned pain modulation; Drug: Placebo Oral Tablet

INTERVENTIONS:
Behavioral: Hypnosis — Hypnosis is a therapeutic method in which the experimenter or therapist make suggestions to individuals after they have undergone a hypnotic induction. This induction is a relaxation procedure designed to focus one's mind and to induce a hypnotic trance in individuals. The hypnotic trance consists in a state of deep absorption, concentration and altered sensations, cognitions and behaviors. Hypnosis can be used for pain control in experimental and clinical settings. In this study, standardized hypnosis including a relaxation technique for the hypnotic induction and a direct hypnotic analgesia technique for the hypnotic suggestions will be used.
  Other Names: Hypnotic suggestions
Behavioral: Meditation — Meditation is a relaxation method that can be used to reduce pain symptoms and pain perception in clinical and experimental situations. In this study, a standardized mindfulness meditation session of 20 minutes will be used to induce a relaxation and an analgesic effect in participants. Mindfulness meditation is a practice intended to increase mindfulness and awareness of the self and the environment by techniques of controlled breathing, focus on neutral elements, and observation of one's thoughts and emotions without judgment.
  Other Names: Mindfulness meditation
Other: Conditioned pain modulation — Conditioned pain modulation (CPM) is a pain inhibition mechanism that is used to assess endogenous analgesia capacity. The method to evaluate CPM in healthy individuals and patients with pain includes both a conditioning stimulus (a noxious stimulus that induces CPM) and a test stimulus (a noxious stimulus used to evaluate the analgesic response to the conditioning stimulus). In this study, the conditioning stimulus will be a cold pressor test (two-minutes immersion of one hand in ice water) and the test stimulus will be a two-minutes thermal noxious stimulus delivered by a contact thermode.
  Other Names: CPM; Pain modulation; Diffuse noxious inhibitory control; DNIC; Hetero-segmental counter-irritation
Drug: Placebo Oral Tablet — A placebo is a substance (or treatment) with no active therapeutic effect. The placebo effect (analgesia) in this study will be induced by the oral administration of one inert tablet (sugar pill). The tablet is a round, hard, white, flat-faced tablet with no active ingredient. The participant is told that the tablet is an active drug, more specifically an analgesic or a painkiller, that is used to achieve analgesia, relief from pain. This placebo condition is used to induce a diffuse analgesic effect in participants.
  Other Names: Placebo analgesia; Placebo effect; Placebo

SUMMARY:
Introduction: Many interventions such as hypnosis, mindfulness meditation, conditioned pain modulation and placebos have been shown to effectively reduce pain both in the laboratory and in clinical settings. However, little is known about their neurophysiological mechanisms of action. Analgesia induced by these techniques is thought to be based on opioidergic and non-opioidergic mechanisms (potentially endocannabinoid mechanisms). Objective: Our main objective is to evaluate the effect of hypnosis, meditation, conditioned pain modulation and placebo on blood concentrations of endocannabinoids (anandamide, 2-arachidonylglycerol, N-palmitoyl-ethanolamine, N-oleoylethanolamide), endogenous opioids (β-endorphins, met / leu-enkephalins, and dynorphins) and norepinephrine in healthy adults. Methods: This study is based on a single-group pre-experimental research design in which two experimental sessions including hypnosis or meditation, conditioned pain modulation and placebo interventions will be completed by all participants. In order to have a better description of the sociodemographic and clinical characteristics of the sample, information will be collected by questionnaires or tests filled by participants at baseline, including: age, sex, language, culture, religion, salary, menstrual cycle of women, medication (if any), mood, anxiety, pain catastrophizing, mindfulness, hypnotic susceptibility, and DNA information. Outcome measures will be collected before, during and after each intervention. The primary outcome is plasma concentrations of endocannabinoids. Secondary measurements include plasma concentrations of endogenous opioids and norepinephrine; change in pain intensity during the thermal noxious stimuli; and autonomic nervous system variability (as measured by heart rate variability). Anticipated results: The investigators expect a positive relationship between the change in pain intensity (analgesia) induced by the interventions (hypnosis, meditation, conditioned pain modulation, and placebo) and the change (increase) in plasma concentrations of endocannabinoids, opioids, and norepinephrine in healthy adults. It is also believed that the interventions will influence heart rate variability. Moreover, it is expected that there will be a relationship between the efficiency of the analgesic intervention and some gene polymorphisms associated to pain modulation and endocannabinoids, opioids or norepinephrine in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Being an healthy adult aged 18-45 years old with no prior experience of hypnosis.

Exclusion Criteria:

* Having difficulty understanding french language
* Having a vulnerability to dissociative or psychotic episodes
* Having a diagnosed medical condition or diagnosis of chronic pain leading to kidney, liver, dermatological, respiratory, hematological, immunological, cardiovascular, inflammatory, rheumatologic, endocrine, metabolic, neurological or psychiatric pathologies
* Being pregnant or breast-feeding
* Having a body mass index over 40
* Using medication, recreational drugs or other agents that affect the central nervous system or the perception of pain (e.g., analgesics, opioids, antiepileptics, muscle relaxers)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline concentration of endocannabinoids at the end of the intervention | Immediately before and after each intervention
  Concentrations (ng/ml) of endocannabinoids (anandamide, 2-arachidonylglycerol, N-palmitoyl-ethanolamine, N-oleoylethanolamide) will be measured in the plasma of participants

SECONDARY OUTCOMES:
Change from baseline concentrations of opioids at the end of the intervention | Immediately before and after each intervention
  Concentrations (ng/ml) of opioids (beta-endorphins, met/leu-enkephalins, and dynorphins) will be measured in the plasma of participants
Change from baseline concentrations of norepinephrine at the end of the intervention | Immediately before and after each intervention
  Concentrations (ng/ml) of norepinephrine will be measured in the plasma of participants
Quantitative aspect of pain | Immediately before and after each intervention
  Quantitative aspect of pain, or pain intensity, will be measured and averaged for the entire duration (two minutes) of the pain tests on a Computerized Visual Analog Scale (CoVAS). This CoVAS scale ranges from 0% to 100%. Higher values on this scale represent more intense pain.
Measure of the autonomic nervous system | Immediately before, during and immediately after each intervention
  This outcome will be measured by heart rate variability
DNA in salivary sample | Immediately after all the interventions have been completed, which will be during the second session after the pill has been ingested
  DNA polymorphisms potentially associated with analgesia, endocannabinoids, opioids or norepinephrine

OTHER OUTCOMES:
Anxiety | Immediately before each intervention
  This outcome will be measured on the State-Trait Anxiety Inventory (form Y)
Mood | Immediately after the consent form has been signed, before any intervention is performed
  This outcome will be measured by the Beck Depression Inventory
Pain catastrophizing | Immediately after the consent form has been signed, before any intervention is performed
  This outcome will be measured by the Pain Catastrophizing Scale (PCS). The PCS inquire participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain. Each item of the PCS is scored on a 5-point scale where 0 = not at all and 4 = all the time. PCS yields three subscale scores assessing rumination, magnification and helplessness. The PCS total score is computed by summing responses to all 13 items. The PCS yields a total score ranging from 0 to 52. Higher values on this scale represent a greater tendency of the subject to perceive pain negatively and to foresee the consequences of pain in a more catastrophic way.
Hypnotic susceptibility | Before the hypnosis intervention is performed, during the first session (immediately after the conditioned pain modulation intervention is completed)
  This outcome will be measured by the Stanford Hypnotic Susceptibility Scale: Form A (SHSS:A). This scale was developed to measure susceptibility to hypnosis with items increasing in difficulty. Following a standardized hypnotic induction, the hypnotized individual is given 12 suggestions. Each suggestion is scored on 1 (0 if failed and 1 if passed). SHSS:A yields a total score between 0 and 12. The higher the total score (on 12), the more responsive to hypnosis the subject is.
Hypnotic depth | Immediately after each hypnotic suggestions that will given during the Stanford Hypnotic Susceptibility Scale: Form A and during the hypnosis intervention
  This outcome will be measured by the Long Stanford Scale. Each item (i.e., hypnotic suggestion) is scored on 10 where 0 = wide awake, 1 = borderline, 2 = light, 5 = deep, 10 = very deep. Higher scores suggest greater hypnotic depth for the item (hypnotic suggestion).

CONTACTS AND LOCATIONS:
Overall Officials: Serge Marchand, Ph.D., Principal Investigator — Université de Sherbrooke; Guillaume Leonard, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- CRCHUS: Centre de recherche du centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided